CLINICAL TRIAL: NCT00003670
Title: Phase II Study of LY353381-HC1 Administered to Women With Refractory Ovarian Cancer
Brief Title: Hormone Therapy With Arzoxifene Hydrochloride in Treating Women With Metastatic Refractory Ovarian Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 2145; LILLY-H4Z-MC-JWWJ; MDA-DM-98225; CDR0000066767
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2008-04

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

INTERVENTIONS:
Drug: arzoxifene hydrochloride

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of ovarian cancer cells. Hormone therapy using arzoxifene hydrochloride may fight ovarian or peritoneal cancer by blocking the use of estrogen by the tumor cells.

PURPOSE: This phase II trial is studying how well arzoxifene hydrochloride works in treating women with metastatic refractory ovarian cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate response rate to arzoxifene hydrochloride in patients with metastatic refractory ovarian epithelial cancer or primary peritoneal cancer. II. Determine the time to progressive disease, time to treatment failure, response duration, and survival of these patients. III. Assess the safety of this treatment in these patients. IV. Measure changes in serum estradiol, follicle stimulating hormone, luteinizing hormone, and sex hormone binding globulin during this treatment in these patients.

OUTLINE: Patients receive oral arzoxifene hydrochloride daily at a fixed dose. Treatment continues in the absence of unacceptable toxicity or disease progression.

PROJECTED ACCRUAL: Not specified

National Cancer Institute (NCI) registered this trial with Eli Lilly as sponsor. NCI did not update the record when the trial completed. In June 2012, NCI transferred the trial to Lilly's clinicaltrials.gov account and Lilly updated the record with the trial completion date. This trial is not an applicable trial under Food and Drug Administration Amendments Act of 2007 (FDAAA).

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic refractory ovarian epithelial cancer OR primary peritoneal cancer provided the clinical and pathological features of the tumor are similar to primary ovarian epithelial carcinoma Patients must have received prior chemotherapy including at least one platinum analogue and one taxane analogue unless patient is poor candidate for these treatments due to neuropathy, nephropathy, or hypersensitivity (to Taxol only) Bidimensionally measurable disease by x-ray, CT scan, MRI, or physical exam Ascites not considered measurable or evaluable Hormone receptor status: Estrogen receptor status must be known or tissue must be available for analysis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Sex: Female Menopausal status: Not specified Life expectancy: At least 24 weeks Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL (transfusion-independent) Prothrombin time or activated partial thromboplastin time no greater than 1.25 times upper limit of normal (ULN) Hepatic: Bilirubin no greater than 1.5 times normal ALT or AST no greater than 2.5 times ULN (ALT and AST no greater than 5 times ULN in the presence of liver metastases) Renal: Creatinine no greater than 1.5 ULN Other: No other malignancy within the past 5 years except adequately treated nonmelanomatous cancer of the skin or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No more than 2 prior chemotherapy regimens (including repeated drug combinations) for patients with potentially platinum-sensitive disease No more than 3 prior chemotherapy regimens (including repeated drug combinations) for patients with platinum resistant disease At least 6 weeks since mitomycin or nitrosoureas At least 3 weeks since other prior chemotherapy Recovered from prior chemotherapy Endocrine therapy: At least 3 weeks since hormone replacement therapy No prior hormonal therapy for ovarian cancer Radiotherapy: At least 2 weeks since prior radiotherapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-10; Study Completion 2001-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej P. Kudelka, MD, Study Chair — M.D. Anderson Cancer Center
Locations (4):
- United States (4):
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Abington Memorial Hospital, Abington, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas